CLINICAL TRIAL: NCT00297466
Title: Strategies to Help Adult ED Patients Quit Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA017812
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2006-02

CONDITIONS: Tobacco Use
Keywords: tobacco use; smoking cessation; emergency department
MeSH Terms: conditions — Tobacco Use; Smoking Cessation; Emergencies | interventions — Motivational Interviewing

INTERVENTIONS:
Drug: transdermal nicotine patches
Behavioral: Motivational interview

SUMMARY:
The purpose of this study is to determine whether a brief, focused intervention in the hospital emergency department is effective in helping adults quit smoking.

DETAILED DESCRIPTION:
In urban communities, the prevalence of tobacco use among adults visiting a hospital emergency department (ED) nears 40%, well in excess of the 25% smoking prevalence rate of the general population. Many of these patients lack easy access to primary care, suggesting the ED may be an attractive locus to initiate tobacco cessation efforts. With over 100 million annual visits to U.S. EDs, it may be possible to engage millions of smokers in tobacco cessation efforts. The major purpose of this study is to examine whether a multicomponent intervention delivered in the ED by a Lay Educator to adult smokers interested in quitting is more likely to result in cessation than usual care. A secondary goal is to test whether patients who present to the ED with a tobacco-related illness (as indicated by ICD9 code) are more likely to quit than ED smokers with a non-tobacco-related condition. This will allow us to test the validity of the "teachable moment" as an opportune time to engage patients in considering a behavioral change. The proposed study is a randomized trial of a motivational interview, provision of six weeks' worth of nicotine patches, literature, and post-visit follow-up (Enhanced Care) vs. referral to a cessation clinic (Minimal Care) for ED patients who smoke. Eligibility criteria: age > 21 years, contemplation or preparation stage of change, not admitted to hospital. All patients will undergo a standardized stage of change assessment, and measurements of nicotine dependence and exhaled carbon monoxide. All will receive a cessation fact sheet and referral card to the smoking cessation clinic; the cards of those in the Enhanced Care group will have a specific appointment date and time. The Enhanced Care group will receive a language-appropriate pamphlet discussing smoking cessation. We will record the ICD9 codes associated with each visit. Major outcome measure: cessation within 3 months of the ED visit, stratified by treatment group. Secondary outcome measure: cessation within 3 months of the ED visit, stratified by whether the visit was smoking-related. If smokers receiving Enhanced Care are more likely to quit, then the ED could be considered a new, effective locus for tobacco control, potentially reaching several million smokers. If patients with a smoking-related diagnosis for the ED visit are more likely to quit than those with non-smoking-related ICD9, then this supports the construct of the teachable moment.

ELIGIBILITY:
Inclusion Criteria:

* >= 10 cigarettes smoked daily
* being discharged from the ED
* contemplation or preparation stage of change
* speaks English or Spanish

Exclusion Criteria:

* being admitted to hospital
* too ill to consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
3-month cessation rate

SECONDARY OUTCOMES:
3-month quit attempts,
daily cigarette consumption,
stage of change assessment

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Bernstein, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Bernstein SL, Cooperman N, Jearld S, Moadel A, Bijur P, Gallagher EJ. Predictors of in-person follow-up among subjects in an ED-based smoking cessation trial. Am J Emerg Med. 2012 Nov;30(9):2067-9. doi: 10.1016/j.ajem.2012.06.011. Epub 2012 Sep 20. No abstract available. PMID 23000321
- [Derived] Bernstein SL, Bijur P, Cooperman N, Jearld S, Arnsten JH, Moadel A, Gallagher EJ. A randomized trial of a multicomponent cessation strategy for emergency department smokers. Acad Emerg Med. 2011 Jun;18(6):575-83. doi: 10.1111/j.1553-2712.2011.01097.x. PMID 21676054